CLINICAL TRIAL: NCT05649969
Title: STRONG-PD: Support Through Remote Observation And Nutrition Guidance (STRONG) Program For Cancer Patients With Peritoneal Disease
Brief Title: STRONG Program for Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-22117
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Gastrointestinal Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Referral and Consultation; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- STRONG Program (Experimental): the STRONG program includes consultations with a Moffitt dietician, logging intake of food daily into a food diary with a Fitbit smartphone app, and completing questionnaires.
  Interventions: Behavioral: Consultations with Moffitt Dietician; Behavioral: Daily Food Intake Diary with Fitbit smartphone application; Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Consultations with Moffitt Dietician — Participants will have an initial consultation with a dietician and then biweekly follow-up visits (in person or virtually) for 12 weeks.
Behavioral: Daily Food Intake Diary with Fitbit smartphone application — Participants will keep a daily diary of food intake with a Fitbit smartphone application and wear a Fitbit for 12 weeks
Behavioral: Questionnaires — Participants will complete a questionnaire electronically at baseline and again at week 4, 8, 12 and 16.

SUMMARY:
The purpose of the study is to assess the feasibility and participant satisfaction with the Support through Remote Observation and Nutrition Guidance (STRONG) program. The program provides nutrition support for participants living with gastrointestinal cancer who are receiving chemotherapy and surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Gastrointestinal Cancer diagnosis (e.g., colon cancer, appendiceal cancer)
* Peritoneal disease diagnosis
* Received Cytoreductive Surgery and Heated Intra-Peritoneal Chemotherapy (CRS-HIPEC) for curative intent at Moffitt
* Transitioned to an oral diet post-surgery
* Able to speak and read English
* Able to provide informed consent

Exclusion Criteria:

* Documented or observable psychiatric or neurological disorder that would interfere with study participation (e.g., psychosis, active substance abuse)
* Undergoing concurrent treatment for a secondary primary cancer
* Receipt of parenteral or enteral nutrition after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2025-01-21 (Actual)

PRIMARY OUTCOMES:
Feasibility of the STRONG Program | at 12 weeks
  Feasibility of the Support through Remote Observation and Nutrition Guidance (STRONG) program will be assessed using recruitment and retention rates, along with data completion rates.
Acceptability of the STRONG Program | at 16 weeks
  The Acceptability of the STRONG Program measure uses 4 items to indicate participant satisfaction. The measure uses a scale of 0-5, 0 meaning the participant completely disagrees with the statements regarding intervention satisfaction and 5 indicating complete agreement with the statements regarding intervention satisfaction. The measure score ranges from 0-20 with 20 indicating the highest degree of satisfaction.
Adherence to the STRONG Program | at 16 weeks
  Participant adherence to the Support through Remote Observation and Nutrition Guidance (STRONG) program will be assessed by Fitbit dietary log data and dietician care visit data.
Efficacy of STRONG Program on Treatment Outcomes | at 16 weeks
  Efficacy of STRONG program on treatment outcomes will be measured by reviewing the Electronic Health Record for hospital readmissions and cause of readmission

CONTACTS AND LOCATIONS:
Overall Officials: Amir Alishahi Tabriz, MD, PhD, MPH, Principal Investigator — Moffitt Cancer Center; Ben Powers, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided